CLINICAL TRIAL: NCT05036954
Title: Observational Study on the Efficacy and Tolerance of EYEBRID Lenses
Acronym: EYEBRID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 21-0045
Record Dates: First submitted 2021-06-12; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-07

CONDITIONS: Contact Lens Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- no arm
  Interventions: Device: EyeBrid Excel hybrid lenses

INTERVENTIONS:
Device: EyeBrid Excel hybrid lenses — new lenses

SUMMARY:
Technical advances in lenses are continuous and materials are improved. We provide a prospective longitudinal observational study evaluating the efficacy and safety of new EyeBrid Excel hybrid lenses (LCS) in the treatment of severe ametropia and for patients with corneal irregularities.

This study should include 60 patients for a period of three months. The aim of this work is to assess the improvement in the best corrected visual acuity and the good tolerance of this lens.

ELIGIBILITY:
Inclusion Criteria:

* o Wear rigid lenses and complain about their lenses (discomfort, loss, poor vision) or

  * Wear rigid lenses and have objective intolerances (damage to surfaces related to rigid lenses) or
  * Are new wearers of lenses and presenting a strong ametropia (Strong myopia from -5.00 to -30.00d, strong hyperopia from + 4.50d to + 30.00d, strong astigmatism from 2.50d to 12.00d), with or without presbyopia (Addition of 0.75d to 3.50d)
* Any patient diagnosed with Keratoconus stages 1 to 3.
* Be affiliated to the social security system

Exclusion Criteria:

* Patient with contraindications to wearing contact lenses
* Pregnant or breastfeeding woman
* Any minor or over 80 years old
* Any infection, inflammation or abnormality of the anterior segments
* Progressive ocular disorder of the anterior segments for which the wearing of contact lenses would be discouraged;
* Use of systemic or ocular treatment products for which the wearing of contact lenses would be discouraged;
* History of any herpetic keratitis;
* History of any refractive surgery or any irregular cornea (except in cases where the contact lenses examined may be worn by a subject with an irregular cornea, suffering from keratoconus or having undergone refractive surgery);
* Slit lamp observations of greater than grade 1 gravity;
* Vascularization of the cornea with a penetration greater than 1 mm;
* Case of pathological dry eye;
* When a subject has participated in a clinical trial on contact lenses or contact lens care products within the past 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Contact lens wearers, cohort of 60 patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
tolerance assesment | 3 month
  scale of discomfort when using contact lenses

SECONDARY OUTCOMES:
Improvement of visual acuity | 3 month
  measurement of visual acuity by the ETDRS charts
Assessment and quantification of complications | 3 month
  note the number of abscesses

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided